CLINICAL TRIAL: NCT00425204
Title: A Multi-Center, Open-Label Clinical Trial To Determine The Safety of ABX-EGF As Continued Treatment For Patients Who Have Benefited From and Tolerated Prior ABX-EGF Treatment
Brief Title: Study for Patients Who Have Benefited and Tolerated Prior Panitumumab Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20020375; Abgenix Protocol No. ABX-0311; NCT00081185 (obsolete NCT alias)
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Colorectal Cancer; Non-Small Cell Lung Cancer; Prostate Cancer; Solid Tumors; Advanced Renal Cell Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms | interventions — Panitumumab

ARMS (1):
- Open Label (Experimental): Dose received in previous studies will be rolled over to this study. These regimens include: 2.5 mg/kg weekly; 6.0 mg/kg every 2 weeks; and 9.0 mg/kg every 3 weeks.
  Interventions: Drug: Panitumumab (ABX-EGF)

INTERVENTIONS:
Drug: Panitumumab (ABX-EGF) — Dose received in previous studies will be rolled over to this study. These regimens include: 2.5 mg/kg weekly; 6.0 mg/kg every 2 weeks; and 9.0 mg/kg every 3 weeks.

SUMMARY:
A multi-center, open-label, extended treatment, clinical trial examining the safety of administering multiple does of panitumumab by intravenous (i.v.) infusion to patients who have previously received panitumumab and benefited from treatment

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and sign an IRB approved Informed Consent Form
* Male or female 18 years of age or older
* Female patients who are post menopausal (no menstrual period for a minimum of six months), surgically sterilized, or are using an oral or implanted contraceptive, double barrier birth control, or an intrauterine device (IUD) and have a negative serum pregnancy test upon entry into this study; or male patients willing to use contraception upon enrollment and during the course of the study
* Previously received and tolerated panitumumab treatment on studies 20020374 Part 2 or 20030138/20040116
* Is considered "stable" or "responding" based on the RECIST (20020374 Part 2) or WHO (20040116) criteria, at the final treatment visit of the previous panitumumab clinical trial and the screening visit for this study
* No more than 2 months (60 days) have elapsed since the final treatment visit of the previous panitumumab clinical trial
* Karnofsky score > or = 70%

Exclusion Criteria:

* Brain metastases (20040116 patients are allowed only if controlled and asymptomatic)
* Uncontrolled hypercalcemia (calcium level outside the upper limit of normal; antihypercalcemic treatment is allowed). Exception: Patients in the Motzer Intermediate Risk Group from 20020374 Cohort 2 with uncontrolled high corrected calcium (>10 mg/dl) may be enrolled
* Use of any anti-tumor therapy or investigational drug, other than panitumumab, between the last visit of the previous panitumumab study and the initial visit in this 20020375 study
* Prior treatment with another anti-EGFr agent, other than panitumumab
* Myocardial infarction within 1 year prior to entering the study
* Has other cancer that has been active and required treatment within the past 5 years (basal cell carcinoma or cervical carcinoma in situ are allowed)
* Pregnant or breast feeding female; female of childbearing potential (defined as: post menarche and is biologically capable of becoming pregnant) unwilling to use birth control (as defined in the inclusion criteria) during and for 6 months following treatment
* Male patient unwilling to use birth control (as defined in the inclusion criteria) during and for 1 month following treatment
* Known to be HIV positive
* History of any chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the Investigator may increase the risks associated with study drug administration
* Allergy to the ingredients of the study medication or to Staphylococcus Protein A
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-03; Primary Completion 2007-09 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To provide continued, extended panitumumab treatment to subjects who appeared to have benefited from and tolerated previous panitumumab treatment in Studies 20020374 Part 2 or 20030138 and its extension study, 20040116 | Until disease progression, an AE or withdrawn consent

SECONDARY OUTCOMES:
To assess the safety of multidose administration of panitumumab in subjects who received continued and extended panitumumab treatment | Until disease progression, an AE or withdrawn consent

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_954_AMG_954_20020375.pdf
- See also: FDA-approved Drug Labeling — http://www.vectibix.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com